CLINICAL TRIAL: NCT05132985
Title: Neoadjuvant Icotinib With Chemotherapy for Resectable Stage II-IIIB N2 EGFR Mutation-positive Lung Adenocarcinoma: A Phase II Study
Brief Title: Neoadjuvant Icotinib With Chemotherapy for Epidermal Growth Factor Receptor(EGFR)-Mutated Resectable Lung Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, HongxuLiu, Professor, Liaoning Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIC-0102
Record Dates: First submitted 2021-11-14; First posted 2021-11-24 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: NSCLC; EGF-R Positive Non-Small Cell Lung Cancer
Keywords: NSCLC, EGFR, Icotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib+chemotherapy (Experimental): Neoadjuvant chemotherapy (pemetrexed + carboplatin/cisplatin ) will start within 1-3 days from enrollment at 21-day (+/-3 days) intervals (Q3W) prior to surgery. Before surgery a tumor assessment will be done to exclude evidence of progression. Patients with radiographically stable disease or partial response may be considered for operation.
  Icotinib will be given as a neoadjuvant therapy before surgical resection. The recommended dose of Icotinib is 125mg 1tt(Take 1 tablet 3 times a day) orally.
  Surgery: Surgery must be done within the 3rd to 4th week (+7 days) from day 21 cycle 2 of neoadjuvant treatment.
  Adjuvant treatment: Patients receive additional 2 cycles of platinum-based doublet chemotherapy(Researcher decide) on day 1 with intercalated icotinib (D8-15) every 3 weeks, and continued icotinib for 2 years or until the occurrence of disease relapse, metastasis or unacceptable icotinib or chemotherapy toxicity
  Interventions: Drug: Icotinib; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Icotinib — 125mg 1tt(Take 1 tablet 3 times a day) orally.
  Other Names: Conmana
Drug: Cisplatin — 75 mg/m2 (IV，Q3W)
Drug: Carboplatin — AUC 5 (IV, Q3W)
Drug: Pemetrexed — 500 mg/m2 (IV, Q3W)

SUMMARY:
Icotinib is a first-generation inhibitor of EGFR-tyrosine kinase inhibitor in patients with non-small-cell lung cancer (NSCLC). Here we will evaluate neoadjuvant Icotinib with chemotherapy prior to surgery, in patients with resectable stage II-IIIB N2 EGFR mutation-positive NSCLC. The primary endpoint is centrally assessed major pathological response at the time of resection. Secondary endpoints include pathological complete response, objective response rate, R0 resection rate at the time of resection, disease-free survival, and overall survival. Safety and tolerability will also be assessed.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Male or female, aged ≥18 years and ≤75 years
* Histologically or cytologically documented lung adenocarcinoma with completely resectable disease (Stage II-IIIB N2, according to the 8th edition of the IASLC Staging Manual in Thoracic Oncology)
* Complete surgical resection of the primary NSCLC must be deemed achievable, as assessed by an MDT evaluation
* A tumor which harbors either Ex19del or L858R EGFR-TKI-sensitizing mutations, either alone
* ECOG PS 0/1 at enrollment, with no deterioration over the previous 2 weeks prior to baseline or day of first dosing
* Adequate organ and marrow function as defined by:

  * Hemoglobin: ≥9.0 g/dL
  * Absolute neutrophil count: ≥1.5 × 109/l
  * Platelet count: ≥100 × 109/l
  * Serum bilirubin: ≤1.5 ULN
  * ALT and AST: ≤2.5 × ULN
  * Creatinine clearance: ≥60 ml/min
* Life expectancy of 6 months prior to randomization

Exclusion Criteria:

* Prior treatment with systemic anti-cancer treatment for NSCLC, EGFR-TKI treatment or pre-operative radiotherapy
* EGFR-TKI-sensitizing mutations with T790M
* Mixed small cell and non-small-cell lung cancer histology
* T4 tumors infiltrating the aorta, esophagus and/or heart
* Bulky N2 disease
* Candidates for segmentectomies or wedge resections only
* Medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment or any evidence of clinically active ILD
* Severe or uncontrolled systemic diseases/active infections, history of allogeneic organ transplantation, history of primary immunodeficiency, history of another primary malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response(MPR) | Up to approximately 30 months
  Patients with tumors with ≤10% residual viable cancer cells (identified by routine hematoxylin and eosin staining) in the lung primary tumor after neoadjuvant treatment at the time of resection will be considered to have had an MPR.

SECONDARY OUTCOMES:
Pathological complete response (pCR) | Up to approximately 30 months
  Patients with no residual viable tumor cells in any of the specimens (primary tumors, lymph nodes and margins) will be considered to have had a pCR.
Objective response rate(ORR) | Up to approximately 30 months
  defined as the sum of the complete response plus partial response divided by the total number of included patients.
R0 resection rate | Up to approximately 30 months
  Free resection margins proved microscopically;Systematic nodal dissection in its wider form or, if it is not performed, lobe-specific systematic nodal dissection;There should be no extracapsular extension of tumor in nodes removed separately or those at the margin of the main lung specimen.
  ;The highest mediastinal node that has been removed must be negative.
Disease-free survival(DFS) | Up to approximately 72 months
  DFS will be defined as the time from surgery until the first instance of disease recurrence (local or distant) or death due to any cause, whichever occurs first.
Overall survival(OS) | Up to approximately 72 months
  OS will be defined as the time from randomization until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxu Liu, Doctor, Principal Investigator — Liaoning Cancer Hospital & Institute
Locations (1):
- Liaoning Cancer Hospital & Institute, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NSCLC Meta-analysis Collaborative Group. Preoperative chemotherapy for non-small-cell lung cancer: a systematic review and meta-analysis of individual participant data. Lancet. 2014 May 3;383(9928):1561-71. doi: 10.1016/S0140-6736(13)62159-5. Epub 2014 Feb 25. PMID 24576776
- [Background] Giovannetti E, Lemos C, Tekle C, Smid K, Nannizzi S, Rodriguez JA, Ricciardi S, Danesi R, Giaccone G, Peters GJ. Molecular mechanisms underlying the synergistic interaction of erlotinib, an epidermal growth factor receptor tyrosine kinase inhibitor, with the multitargeted antifolate pemetrexed in non-small-cell lung cancer cells. Mol Pharmacol. 2008 Apr;73(4):1290-300. doi: 10.1124/mol.107.042382. Epub 2008 Jan 10. PMID 18187583
- [Background] La Monica S, Madeddu D, Tiseo M, Vivo V, Galetti M, Cretella D, Bonelli M, Fumarola C, Cavazzoni A, Falco A, Gervasi A, Lagrasta CA, Naldi N, Barocelli E, Ardizzoni A, Quaini F, Petronini PG, Alfieri R. Combination of Gefitinib and Pemetrexed Prevents the Acquisition of TKI Resistance in NSCLC Cell Lines Carrying EGFR-Activating Mutation. J Thorac Oncol. 2016 Jul;11(7):1051-63. doi: 10.1016/j.jtho.2016.03.006. Epub 2016 Mar 19. PMID 27006151
- [Background] Cheng Y, Murakami H, Yang PC, He J, Nakagawa K, Kang JH, Kim JH, Wang X, Enatsu S, Puri T, Orlando M, Yang JC. Randomized Phase II Trial of Gefitinib With and Without Pemetrexed as First-Line Therapy in Patients With Advanced Nonsquamous Non-Small-Cell Lung Cancer With Activating Epidermal Growth Factor Receptor Mutations. J Clin Oncol. 2016 Sep 20;34(27):3258-66. doi: 10.1200/JCO.2016.66.9218. Epub 2016 Aug 9. PMID 27507876
- [Background] Hosomi Y, Morita S, Sugawara S, Kato T, Fukuhara T, Gemma A, Takahashi K, Fujita Y, Harada T, Minato K, Takamura K, Hagiwara K, Kobayashi K, Nukiwa T, Inoue A; North-East Japan Study Group. Gefitinib Alone Versus Gefitinib Plus Chemotherapy for Non-Small-Cell Lung Cancer With Mutated Epidermal Growth Factor Receptor: NEJ009 Study. J Clin Oncol. 2020 Jan 10;38(2):115-123. doi: 10.1200/JCO.19.01488. Epub 2019 Nov 4. PMID 31682542
- [Background] Zhong WZ, Chen KN, Chen C, Gu CD, Wang J, Yang XN, Mao WM, Wang Q, Qiao GB, Cheng Y, Xu L, Wang CL, Chen MW, Kang X, Yan W, Yan HH, Liao RQ, Yang JJ, Zhang XC, Zhou Q, Wu YL. Erlotinib Versus Gemcitabine Plus Cisplatin as Neoadjuvant Treatment of Stage IIIA-N2 EGFR-Mutant Non-Small-Cell Lung Cancer (EMERGING-CTONG 1103): A Randomized Phase II Study. J Clin Oncol. 2019 Sep 1;37(25):2235-2245. doi: 10.1200/JCO.19.00075. Epub 2019 Jun 13. PMID 31194613
- [Result] Goldstraw P, Chansky K, Crowley J, Rami-Porta R, Asamura H, Eberhardt WE, Nicholson AG, Groome P, Mitchell A, Bolejack V; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee Advisory Boards and Participating Institutions. The IASLC Lung Cancer Staging Project: Proposals for Revision of the TNM Stage Groupings in the Forthcoming (Eighth) Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 Jan;11(1):39-51. doi: 10.1016/j.jtho.2015.09.009. PMID 26762738